CLINICAL TRIAL: NCT07367633
Title: A Pragmatic, Multicentre, Adaptive, Prospective, Open-label, Blinded Endpoint Randomized Clinical Trial Assessing the Impact of Head-of-bed Positioning at 0-degrees Versus 30-degrees or More on Functional Recovery Following Endovascular Thrombectomy for Anterior Circulation Large Vessel Occlusion Stroke.
Brief Title: Head of Bed After Ischemic Stroke Thrombectomy (HoBIT)
Acronym: HoBIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HoBIT
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Large Vessel Occlusion; Stroke; Ischemic Stroke
Keywords: head of bed; stroke; large vessel occlusion; endovascular thrombectomy; EVT
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Head of bed position of 0-degrees
  Interventions: Other: Head of bed position of 0-degrees
- Control Arm (Other): Head of bed position of 30-degrees or greater
  Interventions: Other: Head of bed position of 30-degrees or greater

INTERVENTIONS:
Other: Head of bed position of 0-degrees — Flat position with the HoB at 0° elevation for a continuous 24-hour period. Turning to the side (left or right) is permitted, as long as there is no head elevation.
  Other Names: HoB position of 0-degrees
  Arms: Intervention Arm
Other: Head of bed position of 30-degrees or greater — Semi-recumbent position with the HoB to at least 30 degrees for a continuous 24-hour period.
  Head and torso must remain elevated at 30 degrees or higher, using the hospital bed's positioning system.
  Other Names: HoB position of >= 30-degrees; HoB position of greater than or equal to 30-degrees; HoB position of ≥ 30-degrees
  Arms: Control Arm

SUMMARY:
Endovascular thrombectomy (EVT), also known as clot retrieval, is a procedure that improves recovery for people who suffer a stroke by removing blood clots from large blood vessels in the brain. However, half of the patients undergoing EVT to remove the clot from a brain vessel still face lasting disabilities or even die within three months.

The investigators of the HoBIT trial are trying to find out if the position of the head of bed improves recovery in patients who undergo EVT after suffering from a stroke.

The purpose of this study is to establish the benefit of head of bed positioning at 0-degrees compared with 30-degrees or more after EVT for improving functional outcomes in adults that suffer from a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older on the date of randomization
* Endovascular thrombectomy (EVT) for large vessel occlusion (LVO) in the anterior circulation, according to current guidelines and local standards of clinical care. The definition of LVO may include the intracranial segment of the internal carotid artery (ICA), and/ or the M1 segment (proximal, mid, distal) of the middle cerebral artery (M1-MCA), and/ or the proximal M2 segment of the MCA (M2-MCA)
* Capable of giving signed informed consent either independently, or by a legally authorized representative (LAR), or via a deferred consent process approved by the relevant ethics committee, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Mechanical ventilatory support for acute medical condition prior to procedure (i.e. required for reasons other than procedure)
* Symptomatic congestive heart failure, chronic obstructive pulmonary disease, or any other medical condition that would make either HoB position inappropriate for patient care in the judgement of the investigator.
* Any condition, such as but not limited to, agitation/ delirium or severe nausea/ vomiting, that, in the view of the investigator, is expected to significantly impede maintaining the assigned HoB
* Any condition with life expectancy of less than 3 months
* Inability to randomize within 1 hour from the end of the EVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2240 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Functional disability | 90±14 days from randomization
  Functional disability assessed with the modified Rankin Scale (mRS) score.
  Scores:
  0 - No symptoms
  1. - No significant difficulty despite symptoms; able to carry out all usual duties and activities
  2. - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. - Moderate disability; requiring some help, but able to walk without assistance
  4. - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. - Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. - Dead

SECONDARY OUTCOMES:
Absolute difference in NIHSS score | Between randomization and 36±12 hours from randomization
  Absolute difference in the National Institutes of Health Stroke Scale (NIHSS) scores
  Scores:
  0 - No stroke symptoms 1-4 - Minor stroke 5-15 - Moderate stroke 16-20 - Moderate to severe stroke 21-42 - Severe stroke
Early neurological improvement | 36±12 hours from randomization, compared with randomization
  Early neurological improvement, defined as an absolute decrease of the National Institutes of Health Stroke Scale (NIHSS) score by 4 points or more
  Scores:
  0 - No stroke symptoms 1-4 - Minor stroke 5-15 - Moderate stroke 16-20 - Moderate to severe stroke 21-42 - Severe stroke
Functional impairment | Day 7 from randomization or discharge if happens first
  Functional impairment assessed with the Modified Rankin Score (mRS)
  Scores:
  0 - No symptoms
  1. - No significant difficulty despite symptoms; able to carry out all usual duties and activities
  2. - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. - Moderate disability; requiring some help, but able to walk without assistance
  4. - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. - Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. - Dead
Functional independence | Day 7 from randomization or discharge if happens first and 90±14 days from randomization
  Functional independence defined as Modified Rankin Score (mRS) of 2 or less
  Scores:
  0 - No symptoms
  1. - No significant difficulty despite symptoms; able to carry out all usual duties and activities
  2. - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. - Moderate disability; requiring some help, but able to walk without assistance
  4. - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. - Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. - Dead
Quality of life assessment | 90±14 days from randomization
  Quality of life assessed with the EuroQol 5-Dimension 5-Level (EQ-5D-5L) Scores range from 1 (full health) to 0 (dead), with negative values indicating states that are "worse than dead".
Intervention adherence | First 24 hours from randomization
  Adherence to the assigned HoB position for 24 hours from randomization, defined as >80% of total time spent in the assigned HoB
Total time spent | First 24 hours from randomization
  Total time spent in the assigned HoB position
Infarct volume | 24 +/- 12 hours from randomization and 5-7 days from randomization
  Infarct volume on the brain imaging (CT/ MRI) performed as part of standard clinical care

CONTACTS AND LOCATIONS:
Overall Officials: Aristeidis Katsanos, MD, Principal Investigator — Population Health Research Institute; Mike Sharma, MD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada